CLINICAL TRIAL: NCT03455894
Title: Evaluation of the DETECT'CHUTE CLINIBED Smart Carpet for Elderly People Fall Detection
Acronym: CLINIBED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: deficient inclusion
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016_58; 2017-A01910-53 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-02-28; First posted 2018-03-07 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Elderly People
Keywords: Fall detection; Smart carpet; Elderly people

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smart carpet (Experimental)
  Interventions: Device: DETECT'CHUTE CLINIBED

INTERVENTIONS:
Device: DETECT'CHUTE CLINIBED — The DETECT'CHUTE carpets will be positioned at night at the foot of the bed and set in motion by the nursing staff as soon as the elderly person goes to bed for the night. They will be withdrawn the next morning after the resident's rise. Each patient will benefit from the mat for 1 month.

SUMMARY:
DETECT'CHUTE CLINIBED is a smart carpet equipped with several sensors. Positioned at the foot of the bed, this system allows detecting i) patient fall out of the bed and ii) when patient is not back to bed after a certain time. When one of these two events is detected, the system then sends a short message syteme (SMS) and/or an email to the medical staff. The aim of this clinical study is to test the system ability to detect and transmit alarms for both those events.

In this clinical trial, the investigators will therefore test the alarms positive and negative predictive values for both the events.

ELIGIBILITY:
Inclusion Criteria:

* residents of the facility free to get up at night (without a barrier)
* residents may or may not be suffering from Alzheimer's disease or related illness.
* having fallen several times in the last 12 months and / or at risk of falling (time up and go test ≥ 20 seconds).

Exclusion Criteria:

* Subject under tutelage
* use of night barriers or other forms of physical restraint deemed necessary by the physician in charge of the unit care or the patient
* Refusal of the resident's relatives.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

PRIMARY OUTCOMES:
the positive predictive value of alerts | During 30 days
  Evaluation of the positive predictive value of alerts issued by the system. In the event of an alert, caregivers will immediately move to the resident's room to see if the alert has signaled a real fall or no return.

SECONDARY OUTCOMES:
the negative predictive value of alerts | During 30 days
  Measure the negative predictive value of fall and fall alerts.
Time limit of the intervention of nurse | During 30 days
  After each alarm reception (fall or return) the intervention time will be estimated.
  Regular rounds made by caregivers at the usual rhythm, and will see the appearance of a fall not signaled by the carpet.

CONTACTS AND LOCATIONS:
Overall Officials: François Puissieux, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU, Lille, France